CLINICAL TRIAL: NCT00178581
Title: Early Enteral Glutamine Supplement to Enteral Nutrition Support of the Major Torso Trauma Patient: Proposal for a Prospective Randomized Clinical Trial
Brief Title: Enteral Glutamine Supplementation for the Patient With Major Torso Trauma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-05-0144; M01RR002558 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2007-12

CONDITIONS: Trauma; Critical Illness; Shock
Keywords: Trauma; Critical Illness; Shock; Enteral Nutrition; Glutamine
MeSH Terms: conditions — Wounds and Injuries; Critical Illness; Shock | interventions — Glutamine

INTERVENTIONS:
Drug: Glutamine

SUMMARY:
Glutamine is considered a conditionally essential amino acid during critical illness. After severe trauma, glutamine supplementation into the gastrointestinal tract may help maintain bowel function. We hypothesize that for the major torso trauma patient, high dose glutamine given enterally during resuscitation from shock and continued during enteral nutrition support is absorbed, available systemically and preserves gut integrity.

DETAILED DESCRIPTION:
In this prospective, randomized, controlled trial of patients with major torso trauma, high-dose enteral glutamine and enteral nutrition will be given to research subjects while controls will receive isocaloric, isonitrogenous enteral support. Enteral tolerance, bowel integrity and permeability will be evaluated. The systemic appearance of glutamine will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients meeting criteria for shock resuscitation
* Major torso trauma
* Admission to the Shock/Trauma Intensive Care Unit

Exclusion Criteria:

* Age <18 years
* Pregnant
* Expected survival < 24 hours
* Bowel in discontinuity
* Renal failure: baseline serum creatinine>3.0 and/or dialysis
* Admission total bilirubin >10 mg/dl
* History of cirrhosis or cirrhosis apparent on exploratory laparotomy
* Asystole or CPR required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-06; Study Completion 2006-09

PRIMARY OUTCOMES:
Gut function

SECONDARY OUTCOMES:
Systemic appearance of glutamine

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M McQuiggan, MS, RD, CNSD, Principal Investigator — University of Texas Medical School at Houston
Locations (1):
- University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Background] McQuiggan M, Kozar R, Sailors RM, Ahn C, McKinley B, Moore F. Enteral glutamine during active shock resuscitation is safe and enhances tolerance of enteral feeding. JPEN J Parenter Enteral Nutr. 2008 Jan-Feb;32(1):28-35. doi: 10.1177/014860710803200128. PMID 18165444